CLINICAL TRIAL: NCT04144842
Title: A First-in-human, Multicenter, Open-label, Phase 1 Study in Patients With Advanced Solid Malignancies to Evaluate the Safety of Intravenously Administered ATOR-1017
Brief Title: Phase 1 Study in Patients With Advanced Solid Malignancies to Evaluate the Safety of ATOR-1017
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alligator Bioscience AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-19-1017-C-01
Record Dates: First submitted 2019-10-08; First posted 2019-10-30 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2022-08

CONDITIONS: Solid Tumor; Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATOR-1017 (Experimental): ATOR-1017 administered by intravenous infusions every 3 weeks until confirmed progressive disease, clear clinical deterioration, unacceptable toxicity or withdrawal of consent
  Interventions: Biological: ATOR-1017

INTERVENTIONS:
Biological: ATOR-1017 — ATOR-1017 is a human monoclonal antibody targeting 4-1BB (CD137)

SUMMARY:
The aim of the study is to assess the safety and tolerability of increasing doses of ATOR-1017 when administered as repeated intravenous infusions to patients with advanced and/or refractory solid malignancies.

ELIGIBILITY:
Major Inclusion Criteria:

A patient is eligible to be included in the study if all the following criteria apply:

* Has a diagnosis of advanced and/or refractory solid malignancy (histologically or cytologically documented)
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has a minimum of one measurable tumor lesion
* Has acceptable hematologic and clinical chemistry laboratory values

Major Exclusion Criteria:

A patient is excluded if any of the following criteria apply:

* Has not recovered from AEs to at least grade 1 by CTCAE version 5.0 due to prior anti-cancer medications
* Has symptomatic, steroid-dependent or progressive brain metastasis/metastases
* Has a history of another primary malignancy, except for: a) Malignancy treated with curative intent and with no known active disease within 2 years prior to first dose of ATOR-1017, b) Adequately treated non-invasive basal skin cancer or squamous cell skin carcinoma, c) Adequately treated uterine cervical cancer stage 1B or less
* Has an autoimmune disorder requiring immune modulating treatment during the last 2 years
* Receives treatment with systemic immunosuppressant medication (except for inhaled and low dose systemic corticosteroids, i.e. ≤10 mg prednisolone or equivalent per day)
* Is a female patient who is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events (AEs) assessed by Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 | From start of study until 28 days after last dose
  Number of participants with treatment-related AEs assessed by CTCAE v 5.0
Safety and tolerability: Dose-limiting toxicities (DLTs) | From first dose of ATOR-1017 (Day 1) until Day 21
  Number of participants with DLTs

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum observed serum concentration of ATOR-1017 (Cmax) | From start of study until end of study (28-56 days after last dose)
Pharmacokinetics: Time to Cmax | From start of study until end of study (28-56 days after last dose)
Pharmacokinetics: Area under the ATOR-1017 serum concentration-time curve (AUC) | From start of study until end of study (28-56 days after last dose)
Immunogenicity: Anti-drug antibody (ADA) titer in serum | From start of study until end of study (28-56 days after last dose)
  Levels of antibodies to ATOR-1017 will be evaluated
Clinical efficacy: Anti-tumor activity assessed by response evaluation criteria in solid tumors for immune-based therapeutics (iRECIST) | From start of study until end of study (28-56 days after last dose)
  Computed tomography (CT) scans of tumors will be evaluated according to iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Sumeet Ambarkhane, MD, Study Director — Alligator Bioscience AB; Gustav Ullenhag, Dr, Principal Investigator — Department of Oncology, Uppsala University Hospital
Locations (3):
- Sweden (3):
  - Department of Oncology, Skåne University Hospital, Lund
  - Fas 1-enheten, Centrum för Kliniska Cancerstudier, Karolinska Universitetssjukhuset, Solna
  - Department of Oncology, Uppsala University Hospital, Uppsala